CLINICAL TRIAL: NCT05833633
Title: Study of Genotype and Phenotype Characterization and Biomarkers Profile in Duchenne Muscular Dystrophy With Small Mutations
Brief Title: Study of Genotype and Phenotype Characterization in Duchenne Muscular Dystrophy With Small Mutations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Brogna Claudia, Pediatric Neurologist, MD, PhD, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3791
Record Dates: First submitted 2023-03-06; First posted 2023-04-27 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Muscular Dystrophy, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — this includes: modifier genes associated to the Lost of ambulation; RNA study on the dystrophin transcript in urinary stem cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group of DMD patients with different type of small mutations (Group 1): Group of DMD patients with different type of small mutations (15 ambulant or not-ambulant patients)
  Interventions: Diagnostic Test: MUSCLE MAGNETIC RESONANCE IMAGING (MRI)
- Group of DMD patients with non sense mutations in treatment with Traslarna (Group 2): Group of 10 ambulant DMD patients with non sense mutations in treatment with Traslarna (3-[5-(2-fluoro-phenyl)-[1,2,4]oxadiazole-3-yl]-benzoic acid).
  Interventions: Diagnostic Test: MUSCLE MAGNETIC RESONANCE IMAGING (MRI)

INTERVENTIONS:
Diagnostic Test: MUSCLE MAGNETIC RESONANCE IMAGING (MRI) — To assess longitudinally at baseline and 1 year later changes on muscle MRI, genetic test, functional motor and respiratory assessments in the DMD group with different type of small mutations and the DMD group with non sense mutations treated with Atarulen in order to better define natural history of these patients. .
  Other Names: Genetic exams; Functional motor and respiratory assessments

SUMMARY:
Improved standards of care and the regular early use of glucocorticoid treatment have changed the natural history of Duchenne muscular dystrophy (DMD), affecting both survival and time of loss of functional milestones. More recently, there has been increasing evidence of an additional benefit from new therapeutic approaches based on mechanisms targeting specific types of mutation, as Atarulen, authorised in the European Union as Translarna since 31 July 2014 to treat DMD boys with non sense mutations. As there is increasing evidence that specific groups of mutations may have different progression of the disease, it has become mandatory to obtain more detailed long-term information about the patterns of progression related to different genotypes. Natural history of DMD boys carrying deletions has been more studied and less is known about boys carrying small mutations that represent 20% of DMD patients. The aim of this project is to better define the natural history of these patients and to better understand the clinical response to mutation-specific therapies aimed at restoring dystrophin protein production.

DETAILED DESCRIPTION:
In the last years, motor functional assessments have helped to define a better natural history of DMD patients, showing different clustering of disease progression according to the genotype and locus of mutation. Within the spectrum of severity of DMD, variability in phenotype among deletions has been previously reported. However all clinical assessments have the common disadvantage of being dependent on patient collaboration and interaction with the examiner. Therefore, the need to identify new biomarkers as measurable indicators of biologic condition has become important. To date several studies have shown that Magnetic Resonance Imaging (MRI) and spectroscopy provide sensitive markers of muscle pathology and disease progression in both upper and lower limbs of DMD subjects, suggesting MRI as a promising non-invasive candidate biomarker. Muscle MRI has the advantage of being relatively independent of patient collaboration. In previous studies, quantitative thigh muscle MRI values highly correlated with clinical outcome measures and loss of ambulation (LOA) and qualitative assessment scoring showed a direct correlation with the the duration of illness and fibro-fatty changes. More recently, our team found a relation between the functional scores and severe involvement on muscle MRI of upper limb in both ambulant and non-ambulant DMD boys. Furthermore, in the last decades the evidence that the age of LOA varies between DMD individuals carrying mutations abolishing dystrophin expression, has suggested the existence of trans-acting variants in modifier genes. It has been recently reported that some single nucleotide polymorphisms (SNPs) in a few identified genes can be considered as DMD modifiers and responsible for some of the inter-individual variability observed in the clinical disease course. To date, variants in five loci have been associated with variability in human DMD sub-phenotypes: Secreted Phosphoprotein 1 (SPP1), Latent Transforming Growth Factor-Beta Binding Protein 4 (LTBP4), Cluster of differentiation 40 (CD40), alfa-actinin-3 (ACTN3), and Thrombospondin 1 (THBS1). These genes are implicated in several interconnected molecular pathways regulating inflammatory response to muscle damage, regeneration, fibrosis or are more directly implicated in muscle power and sprint performance. Described variants have a regulatory function or alter protein sequence and could delay median LOA by approximately 1 to 2 years. Furthermore, more recently, native urine derived stem cells were demonstrated to express dystrophin transcript and protein (following myoblast determination protein 1 (MyoD) differentiation) in both DMD patients and control group and they could be considered a valid cell tool for either genotype characterization and functional studies on both DMD transcript and dystrophin (DYS) protein. So far, the results of the literature on small mutations report a wide variability of clinical findings and it could be hypothesized that the variable trajectories of progression and the overall severity and loss of important milestones may depend by several factors. One could assume that this finding could be related to the different site of mutations and specific exon involvement or to the type of the aminoacidic changes that could be able to produce different expressions of residual protein with subsequent differences in the severity of phenotypes. These points have not been systematically explored and the use of biomarkers may facilitate to identify distinct phenotypes and their correlation with different genotypes. This project aims to investigate whether specific genotype characterization, functional assessments, muscle MRI could help to establish a better genotype and phenotype characterization in a group of DMD patients carrying small mutations. I hypothesize that these tools alone or combined may help to allow describing the natural history.

ELIGIBILITY:
Inclusion Criteria:

- DMD diagnosis confirming a small mutation genotype.

Exclusion Criteria:

* DMD patient enrolled in other clinical trials using genetic approach
* impossibility to perform MRI without sedation
* presence of severe cognitive or behavioral problems

Ages: 4 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All 25 patients had genetically proven DMD diagnosis with a small mutation genotype; the sample includes both ambulant and non ambulant patients; Ten patients of the 25 are in treatment with Atarulen.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Longitudinal Motor changes in 15 DMD boys with different types of small mutations (Group 1) | 1 year
  To found in a cohort of 15 patients with different types of small mutations at baseline (T0) and 1 year later (T1) some differences in motor functional assessments including the six minute walking test and the Performance of the Upper Limb.
Longitudinal respiratory changes in 15 DMD boys with different types of small mutations (Group 1) | 1 year
  To found in the same cohort of 15 patients with different types of small mutations at baseline (T0) and 1 year later (T1) some differences in respiratory data using the Peak Expiratory Flow percentage predicted.
  ,
Longitudinal Muscle MRI changes in 15 DMD boys with different types of small mutations (Group 1) | 1 year
  To found in the same cohort of 15 patients with different types of small mutations at baseline (T0) and 1 year later (T1) some differences in muscle MRI scores
Longitudinal genetic changes in 15 DMD boys with different types of small mutations (Group 1) | 1 year
  To found in the same cohort of 15 patients (prospective cohort) with different types of small mutations at baseline (T0) and 1 year later (T1) some differences in genetic test (urinary stem cells for MiRNA study).
  Genomic DNA exploring the 5 SNPs associated to the LOA will be collected at T0 only

OTHER OUTCOMES:
Longitudinal Motor changes in 10 ambulant DMD boys carrying non-sense mutations treated with Traslarna (Group 2) | 1 year
  To found in a cohort of 10 ambulant DMD boys carrying non-sense mutations treated with Traslarna at baseline (T0) ad 1 year later (T1) some differences in motor functional assessments including the six minute walking test and the Performance of the Upper Limb
Longitudinal respiratory changes in 10 ambulant DMD boys carrying non-sense mutations treated with Traslarna (Group 2) | 1 year
  To found in the same cohort of 10 ambulant DMD boys carrying non-sense mutations treated with Traslarna at baseline (T0) ad 1 year later (T1) some differences in respiratory data using the Peak Expiratory Flow percentage predicted.
Longitudinal Muscle MRI changes in10 ambulant DMD boys carrying non-sense mutations treated with Traslarna (Group 2) | 1 year
  To found in the same cohort of 10 ambulant DMD boys carrying non-sense mutations treated with Traslarna at baseline (T0) and 1 year later (T1) some differences in muscle MRI scores
Longitudinal genetic changes in10 ambulant DMD boys carrying non-sense mutations treated with Traslarna (Group 2) | 1 year
  To found in the same cohort of 10 ambulant DMD boys carrying non-sense mutations treated with Traslarna some differences in genetic test (urinary stem cells for MiRNA study).
  Genomic DNA exploring the 5 SNPs associated to the LOA will be collected at T0 only

CONTACTS AND LOCATIONS:
Overall Officials: CLAUDIA BROGNA, MD, PhD, Principal Investigator — Fondazione Policlinico Gemelli., IRCCS, Rome, Italy
Locations (1):
- Claudia Brogna, Rome, Italy